CLINICAL TRIAL: NCT00034112
Title: Efficacy of Osteopathic Manipulation in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: R21AT000207-01A1 (NIH)
Record Dates: First submitted 2002-04-22; First posted 2002-04-23 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Emphysema
Keywords: chronic obstructive pulmonary disease; combination therapy,; emphysema; exercise; human therapy evaluation; rehabilitation; respiratory disease /disorder therapy; respiratory function; biomechanics; body movement; diaphragm; dyspnea; muscle tension; musculoskeletal system; outcomes research; quality of life; somatic reflex
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive; Motor Activity; Respiratory Aspiration; Dyspnea | interventions — Manipulation, Osteopathic

INTERVENTIONS:
Procedure: osteopathic manipulative treatment

SUMMARY:
The purpose of this study is to determine if osteopathic manipulative treatment (OMT) is effective for persons with emphysema as a component of their chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
OMT sessions are designed to improve chest wall compliance and diaphragmatic function which produce an immediate positive change in pulmonary function parameters and chest wall mobility. This research project will be a significant step in expanding the understanding of the role of OMT in the treatment of chronic lung disease. It is expected to yield evidence that OMT is an important adjunctive modality that improves pulmonary function, increases exercise tolerance, relieves dyspnea, and improves quality of life in those with COPD, and that would have widespread clinical application plus significant economic benefits.

Participants in this study will be randomly assigned to receive either OMT or sham treatments once a week for 13 weeks. Outcome measures will be obtained at baseline; immediately following the first treatment; at 4, 8, and 12 weeks after initiation of treatment; and 4 weeks after termination of the treatment. Outcome variables include pulmonary function tests; quality-of-life questionnaires (including emotional functioning, fatigue, and dyspnea); and measurements of exercise tolerance and chest wall mobility.

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-04; Study Completion 2002-03

CONTACTS AND LOCATIONS:
Overall Officials: Donald R. Noll, Principal Investigator — Kirksville College of Osteopathic Medicine
Locations (1):
- Kirksville College of Osteopathic Medicine, Kirksville, Missouri, United States